CLINICAL TRIAL: NCT05964517
Title: The Effects of the Fascial Distortion Model on Pain Intensity, Cervical Posture, and Joint Position Sense in Patients With Tension-type Headache.
Brief Title: Fascial Distortion Model in Tension Type Headache
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Gaziantep (Other)
Responsible Party: Principal Investigator, Ogr Uyesi Tuba MADEN, Assisstanf Profesor, University of Gaziantep
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022/392
Record Dates: First submitted 2023-07-19; First posted 2023-07-28 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Postural; Defect; Tension-Type Headache; Pain, Neck; Craniovertebral; Syndrome; Proprioceptive Disorders
MeSH Terms: conditions — Tension-Type Headache; Neck Pain; Syndrome; Somatosensory Disorders | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Intervention Model Description: Control and study group
  Facial distortion modeling was applied to the study group for 30 minutes, once a week, for 4 weeks. The control group was followed for 4 weeks and the same evaluations were made to the patients twice.
Who Masked: Participant
Masking Description: Participants dont know in which group enrolled.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): The control group refers to patients with tension-type headache who will not be treated. These patients are only evaluated during follow-up.
- Study Group (Active Comparator): Patients with tension-type headache in the study group are treated. Evaluations are made before and after treatment.
  Interventions: Other: Fascial Distortion Model

INTERVENTIONS:
Other: Fascial Distortion Model — Facial Distortion is a manual therapy technique applied by model physiotherapists. It is a deep tissue massage to the fascial tissue.
  Other Names: Manual therapy
  Arms: Study Group

SUMMARY:
Tension-type headache is a headache that starts from the cervical and suboccipital regions, spreads from the back of the head to the parietal, frontal and temporal regions, and is felt in the form of compression, pressure and heaviness.

Increased muscle and fascia tone in the cervical and cranial region, together with active trigger points and factors that trigger pain, cause tension-type headache. Head and neck fascia serves as an important proprioceptive structure in our body. Abnormal inputs from mechanoreceptors and structures around the joint cause deterioration in joint position sense. This study was planned to investigate the effects of the new facial distortion model on pain intensity, cervical posture and joint position sense, unlike the manual techniques used in previous studies in tension-type headache.

DETAILED DESCRIPTION:
This study was planned as a randomized controlled trial to investigate the effect of fascial distortion model on pain severity, cervical posture and joint position sense in patients with tension headache. Individuals with tension-type headache will be divided into control (n=15) and study group (n=15) by simple random method. Fascial distortion modeling will be applied to the study group for a total of 4 weeks, one session a week for 30 minutes. No application was made to the control group. Evaluations will made for all individuals twice, at baseline and after 4 weeks. Pain severity of individuals was evaluated with VAS and McGill-Melzack Pain Scale, cervical posture with Posturescreen Mobile application, joint position sense with laser cursor-assisted angle repetition test.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of tension-type headache,
* the ages of 20-50 years,
* must be headache complaint for at least 6 months,
* Pain is at least 4 on the visual pain scale.

Exclusion Criteria:

* diagnosis of ervical disc herniation,
* diagnosis of sinusitis, migraine and vertigo,
* diagnosis of scoliosis,
* diagnosis of radiculopathy,
* Having a history of surgery Tumor, cyst or similar findings, Having received any physical therapy for the cervical region before, Having any psychological disorder It is the use of any painkillers during the treatment.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-08-07 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
Pain Evaluation | Change from McGill scale at one month
  The McGill Pain Scale will be used to assess the pain of individuals. The questionnaire consists of four different parts. In the first part, in order to determine the localization of pain. In the second part, there are 20 word groups to be marked to determine the nature of the pain. In the fourth part of the scale, the patient is asked to choose appropriate words to determine the severity of pain. The higher the score, the greater the severity of the pain.
Pain Intensity | Change from VAS at one month
  Pain intensity will be evaluated with the Visual analog scale (VAS). VAS consists of a 10 cm long horizontal line. '0' means no pain, '10' means unbearable pain. For evaluation, the patients were asked to mark the level of pain they felt on this line, and the distance to the starting point was measured with a ruler and the severity of the pain was recorded. The higher the score, the greater the severity of the pain.
Cervical Joint Position sense | Change from joint position sense at one month
  Laser cursor assisted angle repetition test will be used to evaluate cervical joint position sense. The patient is positioned to coincide with the origin point of the laser target table. The patient is first asked to aim at the origin of the target pane with his eyes open. The distance from the point where the patient is standing to the origin is measured in cm. As the deviation distance increases, the sense of joint position worsens.
Posture analysis | Change from posture at one month
  Posturescreen mobile (PostureCo Inc., Trinity, FL, USA) application will be used for cervical posture assessment. Posturescreen Mobile (PSM) is a new photographic mobile application for detecting deviations from ideal posture.The validity and reliability study of the (PSM) application was conducted (118). As a reference point, the canthus of the eye, tragus, 7th cervical vertebra, and acromion will be marked on the photograph by the physiotherapist. Craniovertebral angle and shoulder position angle obtained automatically from the application will be recorded. Forward head posture increases with decreasing craniovertebral angle. The increase in shoulder position angle shows that protraction also increases.

CONTACTS AND LOCATIONS:
Locations (1):
- Tuba Maden, Gaziantep, Sahinbey, Turkey (Türkiye)